CLINICAL TRIAL: NCT05713448
Title: Prevalence of Overweight and Obesity in Adult Patients Suffering From Type 1 Diabetes and Its Effect on Treatment and Associated Co-morbidities
Brief Title: Prevalence of Overweight and Obesity in Adult Patients Suffering From Type 1 Diabetes
Acronym: POOT1
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S64223
Record Dates: First submitted 2022-10-12; First posted 2023-02-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes: Individuals with type 1 diabetes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A registry of individuals with type 1 diabetes that visited the Department of Endocrinology of the University Hospitals of Leuven is established. The objective of this registry is to phenotype patients with type 1 diabetes and obesity and their response to treatment with regard to their outcomes

DETAILED DESCRIPTION:
A registry/database is constructed with data of the individuals with type 1 diabetes that visited the Department of Endocrinology of the University Hospitals of Leuven. Data will be obtained from all visits in terms of sociodemographics, disease origin and disease impact including but not limited to glycemic control, medical history, comorbidities, complications, clinical parameters, anthropometric parameters, biochemical blood values, medical therapy, lifestyle, ...

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Type 1 Diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2099-12-29 (Estimated); Study Completion 2099-12-29 (Estimated)

PRIMARY OUTCOMES:
Prevalence of patients with type 1 diabetes and obesity | Up to 100 years
  Prevalence of obesity in type 1 diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Departement Endocrinology, University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No